CLINICAL TRIAL: NCT05085717
Title: Prevention, Access to Rights, Catch-up Vaccination, Treatment of Conditions During Pregnancy and for Children, Acceptability and Determinants of a Male Prenatal Consultation, Including Screening, Catch-up Vaccination and Access to Social Rights, for Fathers Unborn Children at Montreuil Hospital,
Brief Title: Prevention, Access to Rights, Catch-up Vaccination, Treatment of Conditions During Pregnancy and for Children
Acronym: PARTAGE
Status: Completed | Type: Observational
Sponsor: Raincy Montfermeil Hospital Group (Network)
Responsible Party: Sponsor
Other Study IDs: 2020-A03198-31
Record Dates: First submitted 2021-09-27; First posted 2021-10-20 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: HIV Infection
Keywords: HIV; prevention; pregnancy; health
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Insufficient screening and diagnostic delay play a significant role in sustaining the HIV epidemic by France.

Gender inequalities major factors reinforce social inequalities in order to of heterosexual men born abroad the most later diagnosed with HIV infection. Those gender differences are largely due to efficiency antenatal HIV screening, offered to women every pregnancy and widely accepted: a billed HIV serology in the context of pregnancy monitoring was found for 92% pregnant women benefiting from health insurance in 2015 the health of men is not taken into account in prenatal follow-up current French. The maternity hospital drains a population largely immigrant, often precarious The male prenatal consultation exists but it is not organized: it is possible to implement it, provided that the constraints exerted on men are taken into account.

the projet study the feasibility and the implementation processes place of prenatal consultation of future fathers

DETAILED DESCRIPTION:
Insufficient screening and diagnostic delay play a significant role in sustaining the HIV epidemic by France. No significant decline is recorded in heterosexual, whether born in France or abroad. Gender inequalities major factors reinforce social inequalities in order to of heterosexual men born abroad the most later diagnosed with HIV infection. Those gender differences are largely due to efficiency antenatal HIV screening, offered to women every pregnancy and widely accepted: a billed HIV serology in the context of pregnancy monitoring was found for 92% pregnant women benefiting from health insurance in 2015. The arrival of a child could be an opportunity to screening for the future father as well. However, well that a consultation and a biological assessment intended for future fathers are provided for and fully reimbursed by the social security, the health of men is not taken into account in prenatal follow-up current French. The maternity hospital drains a population largely immigrant, often precarious. She puts in contact with the care of pregnant women who were sometimes distant, but not their companions: beyond the issue of reduction of the hidden HIV epidemic, increased needs for prevention and access to health appeared to us for the pilot phase of this project.

ELIGIBILITY:
Inclusion Criteria:

* For future fathers

  * are eligible for a prenatal consultation all adult men living in Ile de France whose companion is followed at the intercommunal hospital of Montreuil for a pregnancy Evolutionary.
  * having expressed no opposition to participation in the research

For future mothers

* all adult women newly enrolled in the maternity ward of the Montreuil intercommunal hospital centre for a progressive pregnancy declaring a partner involved in pregnancy and residing in Ile de France.
* having expressed no opposition to participation in the research

Exclusion Criteria:

* Persons who are unable to give their non-opposition due to a poor understanding of the French language

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population targeted by the data collection is the same as the population targeted by the intervention.
  Are eligible for a prenatal consultation all men living in Ile de France including the companion is followed at the intercommunal hospital of Montreuil for a progressive pregnancy.
  Women are also targeted by data collection. All women are eligible newly enrolled in the maternity ward of the Montreuil intercommunal hospital centre for a progressive pregnancy declaring a partner involved in the pregnancy and residing in Ile de France.
Sampling Method: Non-Probability Sample
Enrollment: 1347 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
evaluation of the proportion of fathers-to-be who fathers who accepted prenatal consultation among | 6 months
  Study the feasibility and processes of setting up the prenatal consultation of future fathers, through the different modalities proposed (in the maternity ward, elsewhere in the hospital, in the heart of city; during the day or in the evening; with or without an appointment) over a period of 26 months at the hospital intercommunal of Montreuil.

SECONDARY OUTCOMES:
impact of male counselling on testing for HIV and other infections | 6 months
  Assessing the impact of male counselling on testing for HIV and other infections
impact of male consultation on vaccination coverage, | 6 months
  Evaluate the impact of male consultation on other interventions: on vaccination coverage, social security coverage and on the declaration of a attending physician.

CONTACTS AND LOCATIONS:
Locations (1):
- Pauline Penot, Montreuil, France

REFERENCES:
- [Background] Piffaretti C, Looten V, Rey S, Fresson J, Fagot-Campagna A, Tuppin P. Management of pregnancy based on healthcare consumption of women who delivered in France in 2015: Contribution of the national health data system (SNDS). J Gynecol Obstet Hum Reprod. 2018 Sep;47(7):299-307. doi: 10.1016/j.jogoh.2018.05.014. Epub 2018 Jun 2. PMID 29870831
- [Background] Kigozi IM, Dobkin LM, Martin JN, Geng EH, Muyindike W, Emenyonu NI, Bangsberg DR, Hahn JA. Late-disease stage at presentation to an HIV clinic in the era of free antiretroviral therapy in Sub-Saharan Africa. J Acquir Immune Defic Syndr. 2009 Oct 1;52(2):280-9. doi: 10.1097/QAI.0b013e3181ab6eab. PMID 19521248
- [Derived] Penot P, Jacob G, Guerizec A, Trevisson C, Letembet VA, Harich R, Phuong T, Renevier B, Manuellan PE, du Lou AD; Partage Study Group. Implementing a prenatal health screening intervention for future fathers in Montreuil, France: most users are immigrants facing hardship. BMC Public Health. 2024 Oct 28;24(1):2982. doi: 10.1186/s12889-024-20388-x. PMID 39468472